CLINICAL TRIAL: NCT04300478
Title: The Effects of Acute Resistance Exercise on Energy Balance Regulation Among Breast Cancer Survivors
Brief Title: Appetite and Exercise in Breast Cancer Survivors
Acronym: EARNESt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado Clinical & Translational Sciences Institute (Other); National Center for Advancing Translational Sciences (NCATS) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-1974.cc; UL1TR002535 (NIH); KL2TR002534 (NIH); TL1TR002533 (NIH); P30CA046934 (NIH)
Record Dates: First submitted 2020-02-25; First posted 2020-03-09 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2023-03

CONDITIONS: Overweight; Breast Cancer; Obesity
Keywords: Appetite; Energy intake; Energy metabolism; Nutrition; Exercise
MeSH Terms: conditions — Overweight; Breast Neoplasms; Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: Individuals will be randomized to either sedentary control/REx or REx/sedentary control in a 1:1 manner using online software (http://www.randomization.com).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sedentary Control/REx (Other): Subjects will complete the Sedentary control testing sessions, have a 7-14 day washout period, and then complete the REx
  Interventions: Behavioral: REx Condition First; Behavioral: Sedentary Control Condition First
- REx/Sedentary Control (Other): Subjects will complete the REx testing sessions, have a 7-14 day washout period, and then complete the Sedentary control
  Interventions: Behavioral: REx Condition First; Behavioral: Sedentary Control Condition First

INTERVENTIONS:
Behavioral: REx Condition First — REx condition: Participants will complete a whole-body REx workout consisting of 1-set to failure (e.g. RPE of 9-10 on 10-point scale on final reps) on 12 exercises in the Exercise Research Laboratory (located in the CTRC), with a 3-minute rest between exercises. Participants will complete the following exercises: leg press; leg extension; leg curl; hip abduction; hip adduction; chest press; overhead press; seated row; overheard pulldowns and assisted triceps dips on Cybex resistance equipment; barbell calf raises on a Smith machine; and dumbbell biceps curls. Resistance for the REx trial will be determined based on the exercise familiarization session. Specifically, we will target a resistance level needed for each participant to complete ~12-15 repetitions per exercise, using proper form, with an RPE of 9-10 on a 10-point scale on final reps. This protocol eliminates the need for max testing in order to set an exercise protocol off of a specific intensity based on % of 1RM.
Behavioral: Sedentary Control Condition First — Sedentary control condition: Participants will sit quietly in a seated position for the entire duration of this condition.

SUMMARY:
The overall aim of this research is to investigate the acute effects of resistance exercise (REx) on the hormonal and behavioral indices of energy balance regulation in breast cancer survivors. This pilot study is designed to provide preliminary data to support future exercise interventions with more comprehensive energy balance profiling.

DETAILED DESCRIPTION:
After screening, eligible and consented participants will complete baseline evaluations of REE, body composition, and subjective questionnaires to assess energy balance. Eligible and interested individuals will attend an exercise familiarization session in the two weeks before the initial study visit. Individuals will then be randomized to either sedentary control/REx or REx/sedentary control in a 1:1. A washout period of approximately 7-14 days will separate testing sessions.

A randomized cross-over short-term study design was chosen to assessment to profile appetite, energy intake, and physical activity in controlled and free-living settings while also reducing participant burden (as opposed to a long-term intervention). Participants will serve as their own controls, thereby circumventing inter-individual variation in physiology that may confound results. It is anticipated that responses to acute exercise will be amplified in chronic interventions and may therefore be used as a basis for generating hypotheses on the regulation of certain energy balance components. The study will end after the completion of 3 days of dietary intake recall and physical activity measurement for the last participant.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age: 18 - 45 years, since older age may impact appetite regulation45-47 and women >45 are more likely to have begun the menopausal transition (estrogen relates to appetite and eating behavior)
* Body mass index [BMI]: 25 - 35 kg/m2. Since body composition and body mass relate to appetite regulation and energy intake, a narrow BMI range should decrease heterogeneity within the results. The BMI range was chosen to represent a population at risk for developing obesity and associated comorbidities, while also excluding individuals with severe obesity (which may plausibly significantly impact energy intake regulation).
* Pre-menopausal before cancer diagnosis and treatment
* <1 hour/week of planned physical activity by self-report in the previous 12 months, since exercise may alter appetite and response to food
* Diagnosis of primary stage I - II estrogen receptor/progesterone receptor-positive (ER/PR+) breast cancer, according to institutional standards.
* All chemotherapy, radiation, and surgery completed at least two weeks (14 days), but less than 6 months prior to registration

Exclusion Criteria:

* Cancer diagnosis in the last 5 years before breast cancer; any site, excluding melanoma
* History of cardiovascular disease or symptoms suggestive of cardiovascular disease: chest pain, shortness of breath at rest or with mild exertion, syncope
* Diabetes mellitus, uncontrolled hypertension (defined as: systolic blood pressure >160 mmHg or diastolic blood pressure >100mmHg, as measured during the screening visit with participants seated quietly), untreated/uncontrolled thyroid disease, or any other medical condition affecting weight or energy metabolism. Participants who are deemed ineligible based upon uncontrolled hypertension criteria will be referred to their primary care physicians for treatment. If this condition become controlled they will be allowed to be re-evaluated for inclusion in the current trial.
* Unable to exercise due to cardiac, pulmonary, neurological, orthopedic reasons.
* Currently smoking and/or nicotine use.
* Treatment with medications known to significantly affect appetite, weight, energy metabolism, EI or energy expenditure in the last 3 months (e.g. appetite suppressants, lithium, stimulants, anti-psychotics, tricyclic antidepressants).
* Corticosteroid use within the last two weeks
* History of surgical procedure for weight loss at any time (e.g. gastroplasty, gastric bypass, gastrectomy or partial gastrectomy, adjustable banding, gastric sleeve); history of extensive bowel resection for other reasons
* Currently pregnant, lactating or less than 6 months post-partum.
* Score of ≥ 2 on the CAGE (cut-annoyed-guilty-eye opener) questionnaire adapted to include drug use
* Score of > 20 on the Eating Attitude Test - 26 (EATS-26), indicative of disordered eating. Participants with a score >20 on the EATS-26 will be referred to their primary care physician for further evaluation.
* Significant food intolerances/allergies that cannot be accommodated by the University of Colorado Hospital Clinical Translational Research Center (CTRC) Metabolic Kitchen.
* Currently participating in any formal weight loss or physical activity programs or clinical trials for weight loss.
* Other medical, psychiatric, or behavioral limitations that may interfere with participation (as determined by study physician, Dr. Marc-Andre Cornier).
* Unable or unwilling to undergo study procedures

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female Sex
Enrollment: 21 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-05 (Actual)

PRIMARY OUTCOMES:
Ghrelin area under the curve (AUC) in response to exercise or control | 2 years
  Ghrelin will be collected through serial IV collection. Each serum sample will be stored at -80C until analysis Radioimmunoassays will be used to determine serum total ghrelin (Milliipore). Total AUC will be calculated with the Trapezoid method, using all time points over the three hours following the control meal.

SECONDARY OUTCOMES:
Peptide-YY (PYY) area under the curve (AUC) in response to exercise or control | 2 years
  PYY will be collected through serial IV collection. Each serum sample will be stored at -80C until analysis Radioimmunoassays will be used to determine PYY (Millipore). Total AUC will be calculated with the Trapezoid method58, using all time points over the three hours following the control meal.
Subjective ratings of hunger in response to exercise or control | 2 years
  Appetite Ratings will be completed using 100 mm visual analogue scale (VAS) questions (hunger, fullness, and desire to eat) at time points described above. Total AUC will be calculated using the Trapezoid method.
Subjective ratings of food-related cravings in response to exercise or control | 2 years
  Subjects will rate 'food appeal', 'food pleasantness', and 'desire to eat' of validated hedonic and non-hedonic food items using the ImageRate software with 0-100mm VAS scales.
Subjective ratings of appeal/desire for hedonic foods in response to exercise or control | 2 years
  Subjects will rate 'food appeal', 'food pleasantness', and 'desire to eat' of validated hedonic and non-hedonic food items using the ImageRate software with 0-100mm VAS scales.
Subjective ratings of satiety in response to exercise or control | 2 years
  Appetite Ratings will be completed using 100 mm visual analogue scale (VAS) questions (hunger, fullness, and desire to eat) at time points described above. Total AUC will be calculated using the Trapezoid method.
Ad libitum absolute and relative energy intake (EI) | 2 years
  Acute ad libitum EI will be measured during the buffet lunch via the weight and measure method by the dietary staff at the CTRC to measure energy and macronutrient intake following the REx and control conditions. The buffet lunch will consist of 15% more food than predicted requirements and the option to get more food as desired.
Free-living energy intake (EI) for three days following each study day | 2 years
  Acute ad libitum EI will be measured during the buffet lunch via the weight and measure method by the dietary staff at the CTRC to measure energy and macronutrient intake following the REx and control conditions. The buffet lunch will consist of 15% more food than predicted requirements and the option to get more food as desired.
Free-living physical activity for three days following each study day | 2 years
  Activity and sedentary behaviors will be measured with ActivPAL accelerometers for 3 days after each study visit
Total step count for three days following each study day | 2 years
  Activity and sedentary behaviors will be measured with ActivPAL accelerometers for 3 days after each study visit
Sedentary time for three days following each study day | 2 years
  Activity and sedentary behaviors will be measured with ActivPAL accelerometers for 3 days after each study visit

OTHER OUTCOMES:
Resting energy expenditure (REE) | 2 years
  REE will be measured for 20-25 minutes after a period of 30 minutes of quiet rest using an indirect calorimeter with ventilated hood (Parvo Medics metabolic cart). This test measures oxygen consumed and carbon dioxide exhaled to calculate REE (in kilocalories/day) using the Weir formula.
Body composition (fat mass[FM]) | 2 years
  Data on participant's FM will be collected using a full body dual X-ray absorptiometry (DEXA; Hologic Delphi-W, Hologic Inc., Bedford, MA). The scanner will be calibrated according to the manufacturer's guidelines. All participants will undergo a pregnancy test before body composition testing. Body composition variables will be expressed in absolute terms and controlling for height (e.g. FM index: FM [kg]/height [m2])
Body composition (Fat-free mass [FFM]) | 2 years
  Data on participant's FFM will be collected using a full body dual X-ray absorptiometry (DEXA; Hologic Delphi-W, Hologic Inc., Bedford, MA). The scanner will be calibrated according to the manufacturer's guidelines. All participants will undergo a pregnancy test before body composition testing. Body composition variables will be expressed in absolute terms and controlling for height (e.g. FFM will also be expressed in relation to FM (FM:FFM).
Gonadal hormones (estradiol and progesterone) | 2 years
  Additional blood for a single assessment of estradiol (Beckman Coulter) and progesterone (Beckman Coulter) will be collected at baseline during the first study visit to control for these hormones in the statistical analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Ed Melanson, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Univeristy of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Colorado Cancer Center, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Purcell SA, Melanson EL, Afghahi A, Borges VF, Sinelli I, Cornier MA. The effects of resistance exercise on appetite sensations, appetite related hormones and energy intake in hormone receptor-positive breast cancer survivors. Appetite. 2023 Mar 1;182:106426. doi: 10.1016/j.appet.2022.106426. Epub 2022 Dec 17. PMID 36539160
- See also: Main results of the study — https://pubmed.ncbi.nlm.nih.gov/36539160/